CLINICAL TRIAL: NCT04839497
Title: A Phase 2 Multicenter Randomized Single Arm Crossover Trial Evaluating the Safety and Efficacy of Autologous Volar Fibroblast Injection Into the Terminal Limb of Amputees
Brief Title: Multicenter Trial Evaluating the Safety and Efficacy of Autologous Volar Fibroblast Injection Into the Terminal Limb of Amputees.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH1820055
Record Dates: First submitted 2021-03-23; First posted 2021-04-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Amputation

STUDY DESIGN:
Intervention Model Description: Cross over design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Volar Fibroblast Treatment (Experimental): Volar fibroblasts are injected into the residual limb of transtibial amputees
  Interventions: Combination Product: Autologous Volar Fibroblast Injection into the Terminal Limb of Amputees
- Cryoprotectant (No Intervention): Vehicle Control. Interdermal injection of cryoprotectant

INTERVENTIONS:
Combination Product: Autologous Volar Fibroblast Injection into the Terminal Limb of Amputees — Autologous Volar Fibroblasts Treatment- harvested from patient's biopsied volar skin. Intradermal injection of Volar fibroblasts in the residual limb of transtibial amputees.
  Other Names: Autologous Volar Fibroblast Treatment
  Arms: Volar Fibroblast Treatment

SUMMARY:
The study will enroll 20 adults ages 18-75 with a transtibial amputation with mature residual limbs who are ambulatory prosthesis users. Participants will be randomized to either treatment with low dose volar fibroblast injections (n=10) or to vehicle control (n=10). Participants will undergo a biopsy to harvest volar skin for fibroblast expansion and tattooing to identify injection sites on the residual limb. Fibroblasts will be processed at the Hopkins Cellular Therapy Core Lab and volar cells primed for injection will be sent to participating centers for administration. Participants randomized to the treatment group will be treated with low-dose cells. Injections will be administered on at least 1 and up to three separate days over the course of one week. Participants randomized to the vehicle control group will receive injection of cryoprotectant. All participants will be followed at 2 weeks, 1, 2, and 3 months after the last injection. These visits will include a clinical evaluation for complications, non-invasive assessments of skin firmness and thickness, skin appearance, and patient-reported outcomes. After the final monitoring visit, individuals randomized to the vehicle control group will have the opportunity to receive the volar fibroblast injections and will be followed for an additional 3 months.

The investigators hypothesize that (1) There will be no difference in the rate of serious adverse events among patients treated with volar fibroblast injections compared with patients treated with vehicle control, and (2) Patients treated with volar fibroblast injections will have firmer skin on the residual limb compared with patients tread with vehicle alone.

ELIGIBILITY:
Inclusion criteria:

1. Ages 18 to 75, inclusive
2. Must have a transtibial amputation
3. Must be using a prosthesis within the vicinity of 3 months or have had osteo-integration of a prosthetic in place for 1 month
4. In the opinion of the investigator, must be medically able to undergo the administration of study material determined by laboratory tests obtained up to 14 days before baseline for which the investigator identified no clinically significant abnormality.
5. Able to provide written informed consent
6. Females of childbearing potential must: have a negative pregnancy test at screening agree to not become pregnant or breastfeed for the period of the study through 1 month after completion of the study be willing to use a reliable form of contraception during the study.
7. Has healthy skin on the residual limb and is free of severe and active skin disease (excluding those on the residual limb) such as extreme and active eczema or psoriasis, active non-healing wounds, lichen planus, a history of keloid scare formation or lupus as determined by the investigator or study nurse.
8. Willing and able to comply with the scheduled visits, biopsy/injection procedures, wound care instructions treatment plan, and other study procedures for the duration of the study.

Exclusion criteria:

1. A skin erosion deeper than the skin dermis.
2. Ulcers exceeding 4cm in diameter or 2cm in radius
3. Non circular ulcers that cannot tolerate a 1cm margin at all sides
4. Having received any investigational drug within 30 days prior to study entry
5. An allergy history to any study materials including local anesthetic, dimethyl sulfoxide, human albumin, or bovine constituents, hetastarch, or EMLA (lidocaine 2.5% and prilocaine 2.5%).
6. Pregnant, lactating, or trying to become pregnant
7. A history of keloid formation
8. Having a significant medical history that the investigator feels is not safe for study participation (for example, some forms of autoimmune conditions, metastatic cancer, infectious diseases such as HIV, HTLV I/II, Hepatitis B, Hepatitis C).
9. Autoimmune diseases affecting the skin such as lupus.
10. Presence of necrotic ischemic tissue on any stump ulcers, and/or capillary refill on stump skin of greater than 3 seconds
11. Active infection of the residual limb (e.g. osteomyelitis, wound or skin condition with surrounding swelling, erythema, drainage, pain, gangrenous tissue or fever).
12. Active smoker during the study (this includes e cigarettes and any type of tobacco use)
13. We will also exclude those who are on chronic immunosuppressive therapies such as oral steroids, but also those on chronic topical steroids in the area of investigation.
14. Amputees with symptomatic neuromas of the terminal limb within the last 3 months.
15. Known bleeding disorder.
16. Have a history of congenital or idiopathic methemoglobinemia, glucose-6-phosphate deficiencies, or use of medications associated with drug-induced methemoglobinemia. (specifically: Sulfonamides, Acetaminophen, Acetanilid, Aniline dyes, Benzocaine, Chloroquine, Dapsone, Naphthalene, Nitrates and Nitrites, Nitrofurantoin, Nitroglycerin, Nitroprusside, Pamaquine, Paraaminosalicylic acid, Phenacetin, Phenobarbital, Phenytoin, Primaquine, or Quinine.)
17. Quadriplegics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety assessment of complications and adverse events associated with Volar Fibroblast injections | 3 months from the injection visit
  Safety will be evaluated by routinely assessing all complications at each study visit.
  Minor and expected complications may include local injection reactions like bruising and erythema, swelling and pain.
  Minor complications that are not expected include local small hemorrhage (x<1mL), edema, nodules, papules, irritation, dermatitis, pruritus, and cellulitis.
  Serious Adverse Events are defined as unexpected AND serious AND related or possibly related to the study treatment. These may include but are not limited to osteomyelitis.
Efficacy of autologous volar fibroblasts for increasing skin firmness in individuals with a transtibial amputation. | Baseline through 3 months from the injection visit
  Efficacy will be determined by treatment group difference in the pre- post-change in skin firmness at three months post injection. Skin firmness is the level of resistance as measured by a non-invasive hand-held durometer

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Study results will be published and disseminated in accordance with the METRC publication and data sharing policy guide

DOCUMENTS (1):
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT04839497/ICF_000.pdf